CLINICAL TRIAL: NCT02540330
Title: An Open Label, Phase 2 Pharmacokinetic Study of Pre-Surgical Intramuscular and Intraductal Fulvestrant in Women With Invasive Breast Cancer or DCIS Undergoing Mastectomy or Lumpectomy
Brief Title: A Pre-Surgical PK Study of IM and Intraductally Delivered Fulvestrant
Acronym: 007
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision (See Detailed Description)
Sponsor: Atossa Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATOS-2015-007
Record Dates: First submitted 2015-08-28; First posted 2015-09-03 (Estimated); Results first posted 2022-04-05 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Female Breast Carcinoma; Female Ductal Carcinoma In Situ
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intramuscular Fulvestrant (Active Comparator): 500mg fulvestrant administered intramuscularly
  Interventions: Drug: Fulvestrant
- Intraductal Fulvestrant (Experimental): up to 500mg fulvestrant administered intraductally
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant
  Other Names: Faslodex

SUMMARY:
This is an open-label, non-randomized pharmacokinetic study of fulvestrant in women scheduled for mastectomy or lumpectomy. Eligible subjects will be identified with breast cancer or DCIS. The first subject of each of five groups will receive fulvestrant intramuscularly. The subsequent 5 subjects of each group will receive fulvestrant by intraductal instillation. All subjects will be monitored for systemic and local adverse events during the procedure, and following the procedure until mastectomy or lumpectomy. Subjects that receive fulvestrant will undergo serial blood draws to determine fulvestrant blood concentration levels.

DETAILED DESCRIPTION:
This is an open-label, non-randomized pharmacokinetic study of pre-surgical fulvestrant in women scheduled for mastectomy or lumpectomy. Eligible subjects will be identified upon admission to the institution for surgical management of breast cancer or DCIS, specifically mastectomy or lumpectomy. There will be 5 groups, each consisting of 6 subjects. The first subject of each group will receive fulvestrant administered intramuscularly and the next 5 subjects will receive fulvestrant intraductally. Subjects where at least 1 suitable duct is identified may undergo nipple aspiration in order to facilitate duct identification and intraductal infusion of a fulvestrant accompanied by imaging (saline+ ultrasound). A maximum of 5 ducts will receive intraductal infusion of fulvestrant. Across all ducts, the total dose will not exceed 500 mg (10 mL). All subjects will be monitored for systemic and local adverse events during the procedure, immediately following the procedure, within 30 minutes, 1 hour, 4 hours and by phone following discharge on Days +1 and +2, +7, and pre-operative. Subsequent to mastectomy or lumpectomy, subjects will be assessed for systemic adverse events until discharge. Subjects that receive fulvestrant will undergo serial blood draws to determine fulvestrant blood concentration levels.

This study was terminated due to revised commercial analyses including a review of the potential to enroll in a timely manner the planned number of patients. This study was not terminated because of safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 18 years of age or older
3. Scheduled to undergo non-nipple sparing mastectomy for Invasive Breast Cancer or DCIS
4. Pathological diagnosis of Invasive Ductal Breast Cancer or Ductal Carcinoma in Situ requiring mastectomy or lumpectomy
5. Estrogen Receptor-positive pathology
6. ECOG performance scale of 0-1
7. Adequate organ function as defined by the following criteria:

   * Absolute neutrophil count (ANC) ≥ 1500/μl
   * Platelets ≥ 100,000/μl
   * Hemoglobin ≥ 9.0 g/dl
   * Creatinine ≤ 2 times upper limit of normal
   * Bilirubin ≤ 2 times upper limit of normal
   * Transaminases (AST/SGOT and ALT/SGPT) ≤ 2.5 times upper limit of normal
8. Able to sign informed consent
9. Willing to use effective contraception for at least 100 days post study drug administration.

Exclusion Criteria:

1. Concurrent treatment with another anti-estrogen
2. Presence of an active infection requiring systemic therapy
3. The following conditions contra-indicating fulvestrant administration:

   1. Subjects with bleeding diatheses, thrombocytopenia or current anticoagulant use (excluding aspirin and anti-inflammatories)
   2. Subjects with a known hypersensitivity to fulvestrant or any of its formulation components including castor oil, alcohol, benzyl alcohol, and benzyl benzoate.
   3. Severe hepatic impairment.
4. Prior surgery on the ipsilateral breast which interrupts communication of the ductal systems with the nipple
5. Prior radiation to the breast
6. Pregnant or lactating
7. Impaired cardiac function or history of cardiac problems of NYHA Class 111 and IV
8. Poor nutritional state as indicated by a BMI below 20.
9. Presence of serious infection not controlled with systemic therapy
10. History of allergies to Lidocaine or Novocain
11. Concurrent participation in an experimental drug study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Quay, Study Chair — Atossa Therapeutics, Inc.
Locations (3):
- United States (3):
  - The Johns Hopkins School of Medicine, Baltimore, Maryland
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intramuscular Fulvestrant: 500mg fulvestrant administered intramuscularly
  Fulvestrant
- Intraductal Fulvestrant: up to 500mg fulvestrant administered intraductally
  Fulvestrant
Period: Overall Study
Arm/Group | Intramuscular Fulvestrant | Intraductal Fulvestrant
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intramuscular Fulvestrant | Intraductal Fulvestrant | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 67 [59 to 75] | 45 [45 to 45] | 60 [45 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Two Delivery Methods
Description: Number of adverse events per CTCAE v4.0 after treatment with fulvestrant by route of administration
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Intramuscular Route: 500mg fulvestrant
- Intraductal Route: up to 500mg fulvestrant
Arm/Group | Intramuscular Route | Intraductal Route
Number analyzed (Participants) | 2 | 1
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 50 days
Arm/Group | Intramuscular Fulvestrant | Intraductal Fulvestrant
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intramuscular Fulvestrant (N=2) | Intraductal Fulvestrant (N=1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT02540330/Prot_SAP_000.pdf